CLINICAL TRIAL: NCT07331129
Title: Evaluation of Peri-operative Analgesic Efficacy of Ultrasound Guided Transversalis Fascia Plane Block in Cancer Patients Undergoing Inguinal Lymph Node Dissection: A Prospective Randomized Controlled Study
Brief Title: The Analgesic Efficacy of Ultrasound Guided Transversalis Fascia Plane Block in Inguinal Lymph Node Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ayman Sharawy Abdel Rahman Aboul Nasr, Principal investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2510-501-130-203
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Inguinal Lymph Nodes Enlarged
Keywords: transversalis fascia plane block; ultrasound; inguinal lymph node dissection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided transversalis fascia plane block (TFPB). (Active Comparator): Under aseptic precaution, TFPB will be performed under ultrasonographic guidance using a low-frequency convex transducer (Sonosite M turbo, USA). The patient will be placed in the lateral position. The probe will be introduced to orientation just above the iliac crest transversely; and the three abdominal muscle layers will be identified. Then the probe will be moved posteriorly to show the point at which the transversus abdominis muscle and the internal oblique muscle connected into a common fascia, which is just near the quadratus lumborum muscle. A 22-gauge 80-mm block needle will be used just to pierce the transversalis fascia. To confirm the correct needle tip placement, hydro-dissection will be performed using 2 mL of 0.9% saline following a negative check for blood aspiration to be safe from vascular puncture, then 20 ml of 0.25% bupivacaine will be injected. The real-time US scanning confirmed the spread of the LA in the target plane
  Interventions: Procedure: transversalis fascia plane block and surgical sit local anesthetic infiltration
- surgical incision site infiltration with the local anesthetics. (Active Comparator): Patients of this group will receive local anesthetic 20 ml of 0.25% bupivacaine infiltration into the cutaneous and subcutaneous tissues at the surgical site.
  Interventions: Procedure: transversalis fascia plane block and surgical sit local anesthetic infiltration

INTERVENTIONS:
Procedure: transversalis fascia plane block and surgical sit local anesthetic infiltration — inguinal fascial plane block and surgical site local anesthetic infiltration

SUMMARY:
Pain accompanying Inguinal lymph node dissection triggers a complex stress response leading to impairment of pulmonary, immunological and metabolic function. Opioids are the current gold standard drug for postoperative pain relief, however exposure to large doses lead to multiple side effects of varying significance such as nausea, vomiting, dizziness, constipation, respiratory depression, hypoventilation and sleep disordered breathing. Therefore, strategies other than opioids are recommended without sacrificing proper and effective analgesia, especially in cancer patients who are more susceptible to tolerance and addiction.

Transversalis Fascia Plane Block is used in patients undergoing various surgeries like iliac crest bone harvesting, appendicectomy, cecostomy and inguinal hernia repair, often in combination with TAP block. The initial description of TFPB was with patients in the supine position, with a linear array or curvilinear probe placed between the iliac crest and the costal margin. The external oblique, internal oblique and transversus abdominis muscles and the transversus aponeurosis are identified. The entry of the needle has to be in-plane, from the anterior aspect, and after traversing through the deep surface of the transversus abdominis muscle, local anesthetic is injected to separate the transversalis fascia from the transversus muscle. Studies have demonstrated that this intervention blocks the proximal branches of T12 and L1 and to a lesser extent T11 in the plane between the transversus abdominis muscle and the transversalis fascia. Since its initial description, ultrasound (US)-guided TFPB has been explored in many randomized controlled trials for patients undergoing iliac crest bone harvesting, lower segment caesarean section (LSCS), inguinal hernia repair and hip surgeries.

DETAILED DESCRIPTION:
Inguinal lymph node dissection (ILND) is the surgical removal of lymph nodes from the groin. Inguinal lymph node dissection is used to diagnose cancer spread from certain areas (usually penis, vulva, anus or the skin of the legs or torso), remove lymph nodes that may be cancerous or have a high chance of becoming cancerous, reduce the risk that cancer will recure in the future and help providers to determine the options for treatment. ( Pain accompanying ILND triggers a complex biochemical and physiological stress response leading to impairment of pulmonary, immunological and metabolic function. Opioids are the current gold standard drug for postoperative pain relief, however exposure to large doses lead to multiple side effects of varying significance such as nausea, vomiting, dizziness, constipation, respiratory depression, hypoventilation and sleep disordered breathing . Therefore, strategies other than opioids are recommended without sacrificing proper and effective analgesia, especially in cancer patients who are more susceptible to tolerance and addiction.

Ultrasound imaging made the practice of regional anesthesia easier in visualization and identification of usual and unusual position of nerves, blood vessels, needle during its passage through the tissues, as well as deposition and spread of local anesthetics in the desired plane and around the desired nerve . Several abdominal wall blocks are being used by anesthesiologists to provide postoperative analgesia for surgeries involving lower abdominal incisions. Transversus abdominis plane (TAP) block, quadratus lumborum block (QLB) and ilioinguinal-iliohypogastric block (IIIB). Transversalis fascia plane block (TFPB) was first described by Hebbard in the year 2009.

TFPB is used in patients undergoing various surgeries like iliac crest bone harvesting, appendicectomy, cecostomy and inguinal hernia repair, often in combination with TAP block. The initial description of TFPB was with patients in the supine position, with a linear array or curvilinear probe placed between the iliac crest and the costal margin. The external oblique, internal oblique and transversus abdominis muscles and the transversus aponeurosis are identified. The entry of the needle has to be in-plane, from the anterior aspect, and after traversing through the deep surface of the transversus abdominis muscle, local anesthetic is injected to separate the transversalis fascia from the transversus muscle. Studies have demonstrated that this intervention blocks the proximal branches of T12 and L1 and to a lesser extent T11 in the plane between the transversus abdominis muscle and the transversalis fascia. Since its initial description, ultrasound (US)-guided TFPB has been explored in many randomized controlled trials for patients undergoing iliac crest bone harvesting, lower segment caesarean section (LSCS), inguinal hernia repair and hip surgeries.

To our knowledge, there is no randomized controlled study about it until now in cancer patients undergoing inguinal lymph node dissection, so it will be one of the earliest studies that evaluate peri-operative analgesia efficacy of ultrasound guided transversalis fascia plane block in cancer patients undergoing inguinal lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. American society of anesthesiologists (ASA) class I and II.
2. Age ≥ 18 and ≤ 65 Years.
3. Cancer patients for inguinal lymph node dissection.
4. Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.

Exclusion Criteria:

1. Patient refusal.
2. Local infection at the puncture site.
3. Coagulopathies with platelets count below 50,000 or an INR>1.6.
4. Unstable cardiovascular disease.
5. History of psychiatric and cognitive disorders.
6. Patients allergic to medication used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Pain scores using Visual analogue score | 24 hours after the surgery
  Pain scores using Visual analogue score (VAS) (0 mm = no pain to 10mm = worst pain imaginable) at predetermined time intervals (0,1, 2, 4,6, 12 and 24h) postoperative.

SECONDARY OUTCOMES:
Total intra-operative fentanyl consumption | 2-3 hours (Surgery time) surgery
  the rescue analgesia will be administered intra-operative by fentanyl IV and the total fentanyl used will be recorded and compared between the groups
1st time opioids requested post-operative. | 24 hours after the surgery
  In case of postoperative pain recorded, rescue analgesia will be provided as IV morphine (3 mg) then continuous infusion of morphine through Patient Controlled Analgesia ( PCA ) to keep the VAS scores<3. The total 24-hour morphine consumption will be recorded for every patient.
Total post-operative morphine consumption. | 24 hours after the surgery
  The total 24-hour morphine consumption will be recorded for every patient post operative.
Changes and stability in Mean Arterial Blood Pressure (MAP) | every 15 minutes during the surgery then at 1, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Change in Mean Arterial Blood Pressure (MAP) in mmHg
Changes and stability in Heart Rate (HR) | every 15 minutes during the surgery then at 1, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively
  Change in heart rate (HR) in beat\min

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sharawy Abdel Rahman Aboul Nasr, MD, Principal Investigator — National Cancer Institute Cairo University
Locations (1):
- National Cancer Institute Cairo University, Cairo, Egypt